CLINICAL TRIAL: NCT00661193
Title: A Phase II Selection Design of Pharmacodynamic Separation of Carboplatin/Paclitaxel/OSI-774 (Erlotinib; NSC-718781) or OSI-774 Alone in Advanced Non-Small Cell Lung Cancer (NSCLC) Patients With Performance Status 2 (PS-2)
Brief Title: S0709: Erlotinib With or Without Carboplatin and Paclitaxel in Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593575; S0709 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2008-04-17; First posted 2008-04-18 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Erlotinib Hydrochloride; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): Patients receive oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride
- Arm II (Active Comparator): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and oral erlotinib hydrochloride once daily on days 2-16. Treatment repeats every 21 days for 4 courses. Beginning in course 5 and for all subsequent courses, patients receive oral erlotinib hydrochloride alone on days 1-21. Courses with erlotinib hydrochloride repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: erlotinib hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — given IV
  Arms: Arm II
Drug: erlotinib hydrochloride — given orally
Drug: paclitaxel — given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving erlotinib together with carboplatin and paclitaxel may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well erlotinib works when given alone or together with carboplatin and paclitaxel in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To select a regimen (erlotinib hydrochloride with or without carboplatin and paclitaxel) for further testing against standard treatment, based on median progression-free survival for ≥ 3 months, in patients with stage IIIB or IV non-small cell lung cancer with a Zubrod performance status of 2.

Secondary

* To assess the feasibility of selecting patients for a trial based on central EGFR testing of serum in a cooperative group setting.
* To evaluate the objective tumor response rates (confirmed and unconfirmed, complete and partial response), in a subset of patients with measurable disease.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and oral erlotinib hydrochloride once daily on days 2-16. Treatment repeats every 21 days for 4 courses. Beginning in course 5 and for all subsequent courses, patients receive oral erlotinib hydrochloride alone on days 1-21. Courses with erlotinib hydrochloride repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), including any of the following subtypes:

  * Adenocarcinoma
  * Large cell carcinoma
  * Squamous cell carcinoma
  * Unspecified
* Newly diagnosed primary disease OR recurrent disease after prior surgery and/or radiotherapy, meeting 1 of the following staging criteria:

  * Selected stage IIIB disease (T4 [secondary to malignant pleural effusion only], any N, M0)
  * Stage IV disease (any T, any N, M1 [distant metastases present])
* Measurable or nonmeasurable disease by CT scan, MRI, x-ray, physical exam, or nuclear scan

  * The CT scan from a combined PET/CT scan may only be used to document nonmeasurable disease
  * Pleural effusions, ascites, and laboratory parameters are not acceptable as the only evidence of disease
* Shows evidence of EGFR tyrosine kinase inhibitor therapy benefit (i.e., "proteomics positive") prior to study registration
* No untreated brain metastases

  * Patients with treated brain metastases are allowed provided metastases have remained controlled for at least two weeks following treatment, AND patient has no residual neurological dysfunction off corticosteroids
  * Patients with neurologic abnormalities on physical examination or symptoms must have a negative pretreatment CT or MRI scan of the brain 28 days prior to registration

PATIENT CHARACTERISTICS:

* Zubrod performance status 2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 1,000/mm³
* Serum bilirubin normal
* SGOT or SGPT normal
* Serum creatinine ≤ 2 times upper limit of normal OR creatinine clearance ≥ 50 mL/min
* Willing to provide prior smoking history as requested on the prestudy form
* No gastrointestinal (GI) tract disease resulting in an inability to take enteral medication
* No malabsorption syndrome or requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* No significant history of cardiac disease, including any of the following:

  * Uncontrolled high blood pressure
  * Unstable angina
  * Congestive heart failure
  * Myocardial infarction within the past 6 months
  * Cardiac ventricular arrhythmia requiring medication
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy or surgery (thoracic or other major surgery) and recovered
* At least 1 year since prior adjuvant chemotherapy
* No prior systemic hormonal therapy, chemotherapy, or biological therapy for advanced NSCLC
* No prior EGFR inhibitors
* No prior surgical procedures affecting absorption
* No concurrent major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-12; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (124):
- United States (124):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Epic Care - Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute at St. Luke's, Twin Falls, Idaho
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center - Shawnee Mission, Shawnee Mission, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Veterans Affairs Medical Center - Topeka (O'Neil), Topeka, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Randolph Hospital, Asheboro, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Harrington Cancer Center, Amarillo, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib Hydrochloride: Patients receive oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Erlotinib Hydrochloride, Paclitaxel, Carboplatin: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and oral erlotinib hydrochloride once daily on days 2-16. Treatment repeats every 21 days for 4 courses. Beginning in course 5 and for all subsequent courses, patients receive oral erlotinib hydrochloride alone on days 1-21. Courses with erlotinib hydrochloride repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Erlotinib Hydrochloride | Erlotinib Hydrochloride, Paclitaxel, Carboplatin
Started | 33 | 26
Completed | 0 | 0
Not Completed | 33 | 26
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Progression | 27 | 24
Not completed — Not protocol specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib Hydrochloride | Erlotinib Hydrochloride, Paclitaxel, Carboplatin | Total
Number analyzed (Participants) | 33 | 26 | 59
Age, Continuous [Median (Full Range); unit: years] | 74.9 [45.2 to 84.9] | 70.8 [40.9 to 85.9] | 72.4 [40.9 to 85.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 22 | 51
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 3 | 4
  White | 29 | 19 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 27 | 23 | 50
  Squamous | 5 | 2 | 7
  Large Cell | 0 | 1 | 1
  Other | 1 | 0 | 1
Smoking History [Count of Participants; unit: Participants]
  Current | 10 | 9 | 19
  Former | 17 | 11 | 28
  Never | 6 | 6 | 12
Stage [Count of Participants; unit: Participants]
  IIIB | 1 | 1 | 2
  IV | 32 | 25 | 57
Weight Loss Past 6 Months [Count of Participants; unit: Participants]
  <5% | 14 | 16 | 30
  5-<10% | 14 | 7 | 21
  10-20% | 3 | 1 | 4
  >20% | 1 | 1 | 2
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Selection of One of Two Treatment Regimens (Erlotinib Hydrochloride With or Without Carboplatin and Paclitaxel) for Further Study in a Phase III Trial, Based on Median Progression-free Survival for ≥ 3 Months
Time Frame: From date of registration to 3 years or death, whichever comes first
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib Hydrochloride | Erlotinib Hydrochloride, Paclitaxel, Carboplatin
Number analyzed (Participants) | 33 | 26
months | 1.6 [1.4 to 2.3] | 4.6 [3.0 to 6.7]

2. Secondary Outcome: Response Rate (Confirmed and Unconfirmed, Complete and Partial Response) in a Subset of Patients With Measurable Disease
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From date of registration to 3 years or death, whichever comes first
Population: Although 33 patients were eligible for Erlotinib Hydrochloride, only 32 were evaluable for response due to one patient not having measurable disease at baseline.
Measure: Number; unit: participants
Arm/Group | Erlotinib Hydrochloride | Erlotinib Hydrochloride, Paclitaxel, Carboplatin
Number analyzed (Participants) | 32 | 26
participants | 2 | 6

ADVERSE EVENTS:
Time Frame: From date of registration to 3 years or death, whichever comes first.
Description: All SAEs and AEs.
Arm/Group | Erlotinib Hydrochloride | Erlotinib Hydrochloride, Paclitaxel, Carboplatin
Serious Adverse Events (participants affected / at risk) | 10/32 | 7/26
Other Adverse Events (participants affected / at risk) | 32/32 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Hydrochloride (N=32) | Erlotinib Hydrochloride, Paclitaxel, Carboplatin (N=26)
Cardiac General-Other (Cardiac disorders) | 1 | 0
Death not associated with CTCAE term - Death NOS (General disorders) | 3 | 0
Sudden death (General disorders) | 0 | 1
Infection-Other (Infections and infestations) | 1 | 0
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Hydrochloride (N=32) | Erlotinib Hydrochloride, Paclitaxel, Carboplatin (N=26)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Hemoglobin (Blood and lymphatic system disorders) | 11 | 16
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 | 3
Dry eye syndrome (Eye disorders) | 2 | 3
Keratitis (corneal inflammation/ulceration) (Eye disorders) | 2 | 0
Ocular/Visual-Other (Eye disorders) | 2 | 2
Vision-blurred vision (Eye disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 5 | 10
Diarrhea (Gastrointestinal disorders) | 20 | 20
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 2
Gastrointestinal-Other (Gastrointestinal disorders) | 2 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 6 | 3
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 11 | 10
Pain - Abdomen NOS (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 6 | 9
Constitutional Symptoms-Other (General disorders) | 3 | 2
Edema: limb (General disorders) | 5 | 8
Fatigue (asthenia, lethargy, malaise) (General disorders) | 19 | 18
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 0 | 2
Pain - Chest/thorax NOS (General disorders) | 5 | 0
Pain-Other (General disorders) | 3 | 4
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 3
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 1 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1 | 3
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 1 | 2
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 2 | 0
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 | 2
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 2 | 1
Infection-Other (Infections and infestations) | 3 | 2
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 | 4
AST, SGOT (Investigations) | 1 | 3
Alkaline phosphatase (Investigations) | 5 | 6
Bilirubin (hyperbilirubinemia) (Investigations) | 7 | 5
Creatinine (Investigations) | 9 | 5
INR (of prothrombin time) (Investigations) | 1 | 2
Leukocytes (total WBC) (Investigations) | 0 | 8
Lymphopenia (Investigations) | 5 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 8
Platelets (Investigations) | 1 | 7
Weight loss (Investigations) | 12 | 6
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 10 | 7
Anorexia (Metabolism and nutrition disorders) | 12 | 8
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 | 7
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 | 3
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 | 6
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 | 6
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 10 | 8
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 5 | 5
Pain - Back (Musculoskeletal and connective tissue disorders) | 7 | 5
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 3 | 7
Neuropathy: sensory (Nervous system disorders) | 3 | 10
Ocular/Visual-Other (Nervous system disorders) | 2 | 2
Pain - Head/headache (Nervous system disorders) | 2 | 6
Taste alteration (dysgeusia) (Nervous system disorders) | 5 | 7
Tremor (Nervous system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 4 | 3
Mood alteration - anxiety (Psychiatric disorders) | 2 | 3
Mood alteration - depression (Psychiatric disorders) | 1 | 2
Glomerular filtration rate (Renal and urinary disorders) | 3 | 2
Incontinence, urinary (Renal and urinary disorders) | 1 | 2
Pain - Bladder (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Hemorrhage, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 4 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 6
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 7 | 14
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 0 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 | 6
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 21 | 15
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 2
Hemorrhage/Bleeding-Other (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 5 | 6
Thrombosis/thrombus/embolism (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No